CLINICAL TRIAL: NCT04912765
Title: An Open Label, Single-arm, Phase II Neoantigen (NA) Dendritic Cell (DC) Vaccine and Anti-PD1 (Nivolumab) as Adjuvant Treatment in Resected Hepatocellular Carcinoma (HCC) (Group A) and Liver Metastases From Colorectal Cancer (CRLM) (Group B)
Brief Title: Neoantigen Dendritic Cell Vaccine and Nivolumab in HCC and Liver Metastases From CRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7R9
Record Dates: First submitted 2021-05-24; First posted 2021-06-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Colorectal Cancer; Colorectal Carcinoma; Liver Metastases
Keywords: Tumour neoantigens; Tumor neoantigens; Cancer vaccine; Colorectal Cancer; Hepatocellular Cancer; Immunotherapy; anti-PD1
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Colorectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen Dendritic Cell Vaccine and Nivolumab (Experimental): NA DC vaccine every 2 weeks at a dose of 3-5 million cells.
  Adjuvant nivolumab every 2 weeks at 240mg when given concurrently with the vaccine; every 4 weeks at 480mg after vaccine treatment is completed for a total duration of 1 year.
  Interventions: Biological: Neoantigen Dendritic Cell Vaccine; Drug: Nivolumab

INTERVENTIONS:
Biological: Neoantigen Dendritic Cell Vaccine — 10 doses of the vaccine will be administered via intra-dermal injection concurrently with adjuvant nivolumab.
Drug: Nivolumab — 9 doses of 240mg IV nivolumab as a 30 minutes infusion will be administered in combination with NA DC vaccine starting from the second vaccine dose. Upon completion of 10 doses of NA DC vaccine, 480mg IV nivolumab will be administered as a 30 minutes infusion for a maximum of 9 doses.
  Other Names: Opdivo

SUMMARY:
This is a single arm phase II study of adjuvant intra-dermal NA DC vaccine combined with intravenous nivolumab in patients with resectable HCC (group A) or CRLM (group B) planned for curative surgery (with/without local ablation).

DETAILED DESCRIPTION:
Participants will be consented prior to resection of HCC and CRLM. Genomic sequencing of patient's blood and resected tumour will be performed, followed by tumour NA prediction and production. Patients will undergo venesection to generate DCs which will be pulsed with autologous NAs to produce the vaccine. 10 dose of intra-dermal NA DC vaccine will be administered every 2 weeks together with IV nivolumab (starting from the second vaccine dose). Patients will subsequently continue on adjuvant nivolumab to complete 1 year of treatment.

Efficacy will be evaluated based on relapse-free survival (RFS) at 24 months from surgery and the analyses of specific anti-NA immune responses of autologous peripheral T cells by ELISPOT and/or ICS assays. Safety data will also be obtained for patients who have received at least one dose of treatment.

ELIGIBILITY:
Inclusion Criteria:

HCC specific criteria (Group A):

* Participants must have either newly diagnosed or recurrent HCC, confirmed by histology/cytology or clinically by AASLD criteria in cirrhotic subjects amenable for management with curative intent by resection (with or without the addition of local ablation), if they fulfil the following radiological criteria.

  1. Up to three tumours, at least one with a diameter > 3cm
  2. More than three tumours, none with a diameter > 5 cm
  3. Recurrent HCCs are permitted if they were previously treated with curative intent (e.g. by surgery or ablative methods) and with liver-limited recurrence fulfilling criteria (a) and (b)
* Child-Pugh Score 5 or 6
* All participants are required to have imaging studies (CT chest, tri-phasic CT/MRI of the liver, contrast-enhanced CT/MRI of abdomen and pelvis and other suspected/known sites of disease, and bone scans if indicated) confirming no-extra-hepatic metastatic disease within 12 weeks prior to study enrolment.

CRLM specific criteria (Group B):

* Patients with histologically- or cytologically-diagnosed colorectal cancer with liver-limited metastases are eligible to enrol if:

  1. There are no other sites of metastases aside from the liver confirmed by imaging studies (contrast-enhanced CT chest, abdomen and pelvis or contrast-enhanced CT chest and MRI abdomen and pelvis and other suspected sites of disease, and bone scans if indicated) at least 12 weeks prior to study enrolment AND
  2. The liver metastases are amenable and planned for curative surgical resection with or without the addition of local ablation AND
  3. The primary colorectal tumour had previously been resected or is amendable and planned for surgical resection.
* Participants must have received peri-operative chemotherapy or are being planned for adjuvant chemotherapy after curative surgical resection
* Participants with rectal cancer who received neoadjuvant radiation or are planned for adjuvant radiation are allowed into the study.

General Inclusion Criteria:

* Participants are eligible to enroll if they have non-viral related-HCC, or if they have HBV-HCC, or HCV-HCC defined as follows:

  1. Non-HBV non-HCV related HCC
  2. HBV-HCC:

     1. Resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen), OR
     2. Chronic HBV infection as evidenced by detectable HBV surface antigen or HBV DNA. Participants with chronic HBV infection must be on antiviral therapy
  3. HCV-HCC:

     1. Resolved HCV infection as evidenced by detectable antibody, OR
     2. Chronic HCV infection as evidenced by detectable HCV RNA.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Screening laboratory values must meet the following criteria, and should be obtained within 28 days prior to study enrolment:

  1. Adequate hematologic function:

     1. WBC ≥ 2,000/μL (stable, off any growth factor within 4 weeks of study treatment administration);
     2. Neutrophils Absolute ≥ 1,500/μL (stable, off any growth factor within 4 weeks of study treatment administration);
     3. Hemoglobin ≥ 8.5 g/dL (may be transfused to meet this requirement);
     4. Platelet count ≥ 60 × 103/μL (transfusion to achieve this level is not permitted);
  2. Adequate hepatic function:

     1. Serum albumin > 2.8 g/L (transfusion to meet this level is not permitted); and
     2. Serum total bilirubin < 3 mg/dL, and
     3. Serum Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 5 × ULN;
  3. Prothrombin time (PT)-international normalized ratio (INR) < 2.3 or Prothrombin time (PT) < 6 seconds (transfusion to achieve this level is not permitted)
  4. Adequate renal function with a serum creatinine of < 1.5 × ULN or a creatinine clearance > 40 mL/min (Cockcroft-Gault formula)
* Age and Reproductive Status:

  1. Males and females, ages 21 or older.
  2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of study treatment.
  3. Women must not be breastfeeding.
  4. WOCBP must agree to follow instructions for method(s) of contraception (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment.
  5. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment. In addition, male participants must be willing to refrain from sperm donation during this time.
  6. Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, and still must undergo pregnancy testing as described in this section.

Exclusion Criteria:

HCC specific criteria (Group A):

* Target Disease Exceptions

  1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
  2. Any evidence of tumour metastasis or co-existing malignant disease.
  3. Participants showing evidence of macrovascular invasion on imaging tests.
  4. Participants who have undergone a liver transplant or those who are in the waiting list for liver transplantation.
  5. Participants previously receiving any prior systemic therapy, trans-arterial embolization or chemoembolisation (TAE/TACE), selective internal radiation therapy (SIRT) and stereotactic radiation therapy (SBRT) for HCC.

     CRLM specific criteria (Group B)
* Target Disease Exceptions a) Patients with extra-hepatic colorectal metastases.

General Inclusion Criteria:

* Medical Conditions

  1. Active co-infection with:

     1. Both hepatitis B and C as evidenced by detectable HBV surface antigen (HBs Ag) or HBV DNA and HCV RNA, OR
     2. Hepatitis D infection in participants with hepatitis B
  2. Known positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
  3. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the participant to receive protocol therapy, or interfere with the interpretation of study results.
  4. Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
  5. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
  6. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Prior/Concomitant Therapy

  1. Participants receiving or expected to receive IFN-based therapies during the study period.
  2. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
  3. Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to start of therapy.
* Physical and Laboratory Test Findings

  a. Positive pregnancy test
* Allergies and Adverse Drug Reaction

  1. History of severe hypersensitivity to a monoclonal antibody.
  2. History of allergy or hypersensitivity to study drug components
* Other Exclusion Criteria

  1. Prisoners or participants who are involuntarily incarcerated.
  2. Participants who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
24-month Relapse Free Survival | Time from liver resection to first documented disease recurrence or death by any cause, up to 2 years
  To investigate the clinical efficacy of combining NA DC vaccine with nivolumab in resected HCC and resected CRLM patients.
Induced immune response against vaccinated NAs | Time from liver resection to first documented disease recurrence or death by any cause, up to 2 years
  To determine the presence of NA specific T cells in resected HCC and resected CRLM patients after vaccination. Assessed by EPISOT and/or intracellular cytokine staining (ICS) assay with NA peptides in post-vaccination peripheral blood mononuclear cells (PBMC) compared to pre-vaccination PBMCs.

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (AE) | From the time of start of first treatment administered until 100 days after last dose of study treatment
  To determine the safety and tolerability of combining NA DC vaccine and nivolumab
Overall Survival | From time of start of study enrolment to death due to any cause, up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Si Lin Koo, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore